CLINICAL TRIAL: NCT04905459
Title: A Multicenter Study to Evaluate the Performance of Automated Retinal Disease Assessment Software for the Detection of More Than Mild Diabetic Retinopathy
Brief Title: ARDA Software for the Detection of mtmDR
Status: Completed | Type: Observational
Sponsor: Verily Life Sciences LLC (Industry)
Collaborators: Google LLC. (Industry); Optos, PLC (Industry); Nikon Corporation (Unknown); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 101703
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Retinal Imaging and Mydriatic Agents: Subjects will undergo several types of retinal imaging before and after administration of mydriatic agent. Subjects will be administered mydriatic medication to dilate their pupils.
  Interventions: Diagnostic Test: ARDA software application

INTERVENTIONS:
Diagnostic Test: ARDA software application — Subject images will be sent to the investigational ARDA software

SUMMARY:
This is a multicenter, observational study with primary endpoints to determine the sensitivity and specificity of two investigational software devices that detect the presence of more than mild diabetic retinopathy (mtmDR) in healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of Type I or Type II diabetes mellitus:

   meet the criteria established by either the World Health Organization (WHO) or the American Diabetes Association (ADA)
2. Age 22 or older
3. Understand the study and volunteer to sign the informed consent

Exclusion Criteria:

1. Self-reported visual symptoms and persistent blurred vision (greater than 24 hours); including vision loss that cannot be corrected (e.g. with eye glasses).
2. Diagnosed with macular edema, any known retinopathy, radiation retinopathy, or retinal vein occlusion.
3. History of laser treatment of the retina or injections into either eye, or any history of retinal surgery.
4. Scheduled to undergo the following surgeries before completion of the study imaging: cataract surgery (including any related follow-up procedures) or vitrectomy.
5. Currently participating in an interventional study.
6. Participant has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure or glycemic control, microphthalmia or previous enucleation, etc.).
7. Participant is contraindicated for imaging by fundus imaging system used in the study; e.g.

   1. Participant is hypersensitive to light (side effect of medication or due to unknown etiology)
   2. Participant has undergone photodynamic therapy (PDT)
   3. Previous issues with dilation (angle closure, inability to dilate, allergy to dilation drops).
8. Known pregnancy or possibility of pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sites in the U.S.
Sampling Method: Non-Probability Sample
Enrollment: 1012 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Sensitivity of ARDA mtmDR for detection of mtmDR in 45 degree images | 1 day
Specificity of ARDA mtmDR for detection of mtmDR in 45 degree images | 1 day
Sensitivity of ARDA mtmDR for detection of mtmDR in UWF images | 1 day
Specificity of ARDA mtmDR for detection of mtmDR in UWF images | 1 day

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Midwestern University, Glendale, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Catalina Research Institute, Montclair, California
  - Christie Clinic, Champaign, Illinois
  - Northwestern University, Chicago, Illinois
  - MedStar Health Research Institute Baltimore, Baltimore, Maryland
  - Riverside Diabetes Clinic, Riverdale, Maryland
  - Western Michigan University, Kalamazoo, Michigan
  - PMG Research of Winston Salem, Winston-Salem, North Carolina
  - Diabetes & Endocrinology Associates of Stark County, Inc, Canton, Ohio
  - The Heart and Medical Center, P.C, Durant, Oklahoma
  - BMG The Endocrine Clinic, Memphis, Tennessee
  - Clinical Trials Network, Houston, Texas

IPD SHARING:
Plan to Share IPD: No